CLINICAL TRIAL: NCT04327947
Title: Evaluation of Gynecological Acceptability of 3 Health Care Products (Intimate Gel)
Brief Title: Evaluation of Gynecological Acceptability of 3 Health Care Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herbarium Laboratorio Botanico Ltda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: All-S-EP-076888
Record Dates: First submitted 2020-03-26; First posted 2020-03-31 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Atrophic Vaginitis; Vaginal Disease
MeSH Terms: conditions — Atrophic Vaginitis; Vaginal Diseases

STUDY DESIGN:
Intervention Model Description: Clinical trial, triple arm, randomized
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- women, 18-39 y (Experimental): Health volunteers, 18-39 y, with vaginal dryness
  Interventions: Other: Hyaluronic acid - Research product 1; Other: Hyaluronic acid - Research product 2; Other: Hyaluronic acid - Comparator product
- premenopause women (Experimental): Health volunteers, 40 years to premenopause, with vaginal dryness
  Interventions: Other: Hyaluronic acid - Research product 1; Other: Hyaluronic acid - Research product 2; Other: Hyaluronic acid - Comparator product
- climacteric women (Active Comparator): Health volunteers, climacteric, with vaginal dryness
  Interventions: Other: Hyaluronic acid - Research product 1; Other: Hyaluronic acid - Research product 2; Other: Hyaluronic acid - Comparator product

INTERVENTIONS:
Other: Hyaluronic acid - Research product 1 — Health care product (intimate gel)
Other: Hyaluronic acid - Research product 2 — Health care product (intimate gel)
Other: Hyaluronic acid - Comparator product — Health care product (intimate gel)

SUMMARY:
The research was conduct with 3 different products for use in the intimate region in up to 70 research participants, that use the investigational product by 35 ± 2 days. The subjects were follow up throughout the study by a gynecologist for verification of safety, effectiveness and possible adverse events.

DETAILED DESCRIPTION:
At this study, 70 female participants, 18 to 70 years, healthy with complaints of vaginal dryness used the 3 investigational product, each one by 9 days. Between the changes of product use, there were 4 days of wash out. At the 9th day, the participants answered assessment questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Health volunteers
* Non-injured mucosa in the test region;
* Agreement to adhere to study procedures and requirements and attend the institute on the day(s) and time(s) determined for the evaluations;
* Ability to consent to their participation in the study;
* Age from 18 to 70 years old;
* Female participants;
* Vaginal dryness (slight minimum) - according to questions from the gynecologist.

Exclusion Criteria:

* Pregnancy or breastfeeding;
* Skin pathology in the area of application of the product;
* Diabetes Mellitus type 1; insulin-dependent diabetes; presence of complications due to diabetes (retinopathy, nephropathy, neuropathy); presence of diabetes-related dermatoses (plantar ulcer, lipoid necrobiosis, annular granuloma, opportunistic infections); history of episodes of hypoglycemia, diabetic ketoacidosis and/or hyperosmolar coma;
* Current use of the following medications for topical or systemic use:

corticosteroids, immunosuppressants and antihistamines;

* Skin diseases: vitiligo, psoriasis, lupus, atopic dermatitis;
* History of reaction to the category of the tested product;
* Other diseases or medications that may directly interfere with the study or endanger the health of the research participant.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Perceived hydration | 9 days
  Evaluate the perceived hydration, through a subjective questionnaire based on "Standard Guide for Sensory Claim Substantiation"

CONTACTS AND LOCATIONS:
Locations (1):
- Allergisa Pesquisa Dermato-Cosmética Ltda, Campinas, Brazil